CLINICAL TRIAL: NCT02654015
Title: INVEST: A Single Arm, Feasibility Study of Minimally Invasive Endoscopic Surgical Treatment With Apollo for Supratentorial Intracerebral Hemorrhage (ICH)
Brief Title: INVEST Feasibility - Minimally Invasive Endoscopic Surgery With Apollo in Patients With Brain Hemorrhage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: J. Mocco (Other)
Collaborators: MOUNT SINAI HOSPITAL (Other); University at Buffalo (Other)
Responsible Party: Sponsor-Investigator, J. Mocco, Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 16-0027
Record Dates: First submitted 2016-01-11; First posted 2016-01-13 (Estimated); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Intracranial Hemorrhage
Keywords: intracranial hemorrhage; neurosurgery
MeSH Terms: conditions — Intracranial Hemorrhages | interventions — Practice Management, Medical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Medical Management plus Apollo MIES (Experimental): Subjects will receive best medical management for ICH plus they will receive the MIES surgery and use of the Apollo System for clot evacuation.
  Interventions: Device: Apollo MIES; Other: Medical Management

INTERVENTIONS:
Device: Apollo MIES — Subjects will receive best medical management plus MIES (minimally invasive endoscopic surgery with use of the Apollo System.
  Other Names: ICH - Apollo System
Other: Medical Management — Subjects will receive best medical management for intracranial hemorrhage
  Other Names: MM; ICH - Medical Management

SUMMARY:
The primary objective of this multicenter single arm feasibility study is to provide an assessment of enrollment and follow up feasibility for this patient population being treated with the Apollo Minimally Invasive Surgical Treatment (MIES). Patients who do not qualify for the INVEST Feasibility Study will be referred to the INVEST Registry study.

DETAILED DESCRIPTION:
Objective: The primary objective of this multicenter single arm feasibility study is to provide an assessment of enrollment and follow up feasibility for this patient population being treated with the Apollo or Artemis Minimally Invasive Surgical Treatment (MIES). Patients who do not qualify for the INVEST Feasibility Study will be referred to the INVEST Registry study.

Study Design: This study will be a prospective, multi-centered trial that will enroll 50 patients at up to 10 United States (US) centers.

Patient Population: Patients with moderate-large volume (20-80 cc) supratentorial intracerebral hemorrhage (ICH) who present within 24 hours of symptom onset. Enrolled patients will receive minimally invasive endoscopic evacuation with the Apollo system or Artemis Device.

Indication: The Artemis Neuro Evacuation Device is used for the controlled aspiration of tissue and/or fluid during surgery of the Ventricular System or Cerebrum in conjunction with a Penumbra Aspiration Pump. The Penumbra Aspiration Pump is indicated as a vacuum source for the Penumbra Aspiration Systems. The Apollo system has been cleared for the controlled aspiration of soft tissue and/or fluid during endoscopically guided neurosurgery of the ventricular system or cerebrum. In the present study, the researchers propose to investigate the feasibility of studying this patient population for eventual implementation of efficacy trials.

ELIGIBILITY:
Inclusion Criteria:

* Patient age ≥ 22 and ≤ 80, or age < 85 with baseline mRS=0
* Supratentorial ICH of volume ≥ 30 mL < 80 ml (measured using A x B X C/2 method)
* CT/MR demonstrates ICH stability (< 5 cc growth) at 6 hours after admission scan
* If the initial stability scan shows growth, a second stability scan can be performed q12h until stability is demonstrated or until eligibility for the study has lapsed.
* NIHSS ≥ 6
* Presenting GCS 5 - 15
* Historical mRS 0 to 2
* Symptom onset < 24 h prior initial CT
* Apollo MIES can be initiated within 72h of ictus/bleed
* SBP can be controlled < 160 mmHg and sustained at this level for at least 6 hours

Exclusion Criteria:

* Imaging

  * Expanding hemorrhage on stability CT/MR scan
  * "Spot sign" identified on CTA (May perform a second CTA at 12 hours to demonstrate resolution)
  * Hemorrhagic lesion such as a vascular malformation (cavernous malformation, AVM etc), aneurysm, neoplasm
  * Hemorrhagic conversion of an underlying ischemic stroke
  * Infratentorial hemorrhage
  * Large associated intra-ventricular hemorrhage requiring treatment for IVH-related mass effect or shift due to trapped ventricle (EVD for ICP management is allowed)
  * Midbrain extension/involvement
  * Absolute contraindication to CTA, conventional angiography, and MRA
* Coagulation Issues

  * Absolute requirement for long-term anti-coagulation (e.g., Mechanical valve replacement (bio-prostatic valve is permitted), high risk atrial fibrillation)
  * Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency
  * Platelet count < 100 x 103 cells/mm3 or known platelet dysfunction
  * INR > 1.4, elevated prothrombin time or activated partial thromboplastin time (aPTT), which cannot be corrected or otherwise accounted for (i.e., lupus anti-coagulant)
* Patient Factors

  * Presenting GCS 3 or 4.
  * High risk condition for ischemic stroke (high risk Afib (e.g., mitral stenosis with Afib), symptomatic carotid stenosis)
  * Requirement for emergent surgical decompression or uncontrolled ICP after EVD
  * Unable to obtain consent from patient or appropriate surrogate (for patients without competence)
  * Pregnancy, breast-feeding, or positive pregnancy test [either serum or urine] (Woman of child-bearing potential must have a negative pregnancy test prior to the study procedure.)
  * Evidence of active infection [indicated by fever (at or over 100.7 °F) and/or open draining wound] at the time of randomization
  * Any comorbid disease or condition expected to compromise survival or ability to complete follow-up assessments through 180 days.
  * Based on investigator's judgment, patient does not have the necessary mental capacity to participate or is unwilling or unable to comply with protocol follow up appointment schedule.
  * Active drug or alcohol use or dependence that, in the opinion of the site investigator would interfere with adherence to study requirements.
  * Currently participating in another interventional (drug, device, etc) research project.

Ages: 22 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-06-30 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Mocco, MD, MS, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (7):
- United States (7):
  - George Washington University, Washington D.C., District of Columbia
  - University of Louisville, Louisville, Kentucky
  - University of Buffalo, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Geisinger Medical Center, Danville, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Medical Management Plus Apollo MIES: Subjects received best medical management for ICH plus they received the MIES surgery and use of the Apollo System for clot evacuation.
  Apollo MIES: Subjects received best medical management plus MIES (minimally invasive endoscopic surgery with use of the Apollo System.
  Medical Management: Subjects received best medical management for intracranial hemorrhage
Period: Overall Study
Arm/Group | Medical Management Plus Apollo MIES
Started | 50
Completed | 35
Not Completed | 15
Not completed — Death | 12
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 61.5 [38 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 17
  More than one race | 0
  Unknown or Not Reported | 15

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Enrolled Within 730 Days of First Enrollment
Description: Number of participants enrolled within 730 days of first enrollment to determine rate of recruitment
Time Frame: 730 days
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
Participants | 23

2. Primary Outcome: Number of Participants With Available mRS Score
Description: Rate of Successful Follow up Obtainment based on number of participants with available mRS score at 180 days
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
Participants | 47

3. Secondary Outcome: Stroke Impact Scale - Mobility
Description: For each item, the individual is asked to rate the level of difficulty of the item in the past 2 weeks using the following scale:
  * 1 = could not do it at all
  * 2 = very difficult
  * 3 = somewhat difficult
  * 4 = a little difficult
  * 5 = not difficult at all Stroke Impact Scale full scale from 0-45, with higher score indicating better health outcomes
Time Frame: 180 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
score on a scale | 31 [12.5 to 41.5]

4. Secondary Outcome: Stroke Impact Scale - ADLs
Description: For each item, the individual is asked to rate the level of difficulty of the item in the past 2 weeks using the following scale:
  * 1 = could not do it at all
  * 2 = very difficult
  * 3 = somewhat difficult
  * 4 = a little difficult
  * 5 = not difficult at all
  Stroke Impact Scale - ADL's full scale from 0-50, with higher score indicating better health outcomes.
Time Frame: 180 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
score on a scale | 33 [12.5 to 44]

5. Secondary Outcome: EQ-5D-5L
Description: EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L health states, defined by the EQ-5D-5L descriptive system, may be converted into a single index value. scored as 1 = no problem to 5 = severe problem
  Full scale from 0-25, with higher score indicating better health outcomes.
Time Frame: 180 days
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
score on a scale | 12.5 [9.3 to 17.8]

6. Secondary Outcome: Length of Hospital Stay
Description: number of days of hospital stay
Time Frame: average of 14 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
days | 13.5 [7.2 to 22.8]

7. Secondary Outcome: Number of Participants With Modified Rankin Score (mRS) Less Than or Equal to 3
Description: Number of participants with modified Rankin score (mRS) less than or equal to 3 to assess global disability assessed.
  The Modified Rankin Scale (mRS) The scale runs from 0-6, running from perfect health without symptoms to death. 0 - No symptoms.
  1. - No significant disability. Able to carry out all usual activities, despite some symptoms.
  2. - Slight disability. Able to look after own affairs without assistance, but unable to carry out all previous activities.
  3. - Moderate disability. Requires some help, but able to walk unassisted.
  4. - Moderately severe disability. Unable to attend to own bodily needs without assistance, and unable to walk unassisted.
  5. - Severe disability. Requires constant nursing care and attention, bedridden, incontinent.
  6. - Dead.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
Participants | 22

8. Secondary Outcome: Number of Participants Who Meet Both Criteria of Reduction of Hemorrhage Volume
Description: Predominantly or Only ICH: Number of participants who meet both criteria of reduction of reduction to < 15 cc total volume AND >60% reduction in hemorrhage volume on immediate post-treatment CT scan. Number of participants who meet both criteria of reduction of Hemorrhage volume as indication of surgical success.
Time Frame: 180 days
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
Participants | 28

9. Secondary Outcome: Number of Participants With IVH (mGraeb > 0) With an mGraeb Score of Less Than or Equal to 5
Description: Predominantly or Only IVH: number of participants with IVH (mGraeb > 0) with an mGraeb score of less than or equal to 5 on day 7 CT scan. Number of participants with IVH (mGraeb > 0) with an mGraeb score of less than or equal to 5 as indication of surgical success.
Time Frame: Day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
Participants | 19

10. Secondary Outcome: Number of Participants Who Died Within 90 Days of the Procedure
Description: Rate of mortality as Safety Endpoint. Number of participants who died within 90 days of the procedure.
Time Frame: 90 days
Measure: Count of Participants; unit: Participants
Arm/Group | Medical Management Plus Apollo MIES
Number analyzed (Participants) | 50
Participants | 7

ADVERSE EVENTS:
Time Frame: 180 days
Arm/Group | Medical Management Plus Apollo MIES
All-Cause Mortality (participants affected / at risk) | 12/50
Serious Adverse Events (participants affected / at risk) | 24/50
Other Adverse Events (participants affected / at risk) | 25/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medical Management Plus Apollo MIES (N=50)
Altered mental status (Psychiatric disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 1
Chest pain (General disorders) | 1
Hematoma (Blood and lymphatic system disorders) | 1
ICH (Nervous system disorders) | 5
Cardiac arrest (Cardiac disorders) | 3
Pneumonia (Infections and infestations) | 4
Sepsis (Immune system disorders) | 2
Death (General disorders) | 4
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 2
Intraoperative hemorrhage (Surgical and medical procedures) | 1
Postoperative hemorrhage (Surgical and medical procedures) | 1
Cerebral edema (Nervous system disorders) | 2
GI bleed (Gastrointestinal disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
EVD Malfunction (Surgical and medical procedures) | 1
Ventriculitis (Nervous system disorders) | 1
Ventriculostomy Malfunction (Surgical and medical procedures) | 1
Increase lethargy/Encephalopathy (General disorders) | 1
Worsening of hemorrhage edema and midline shift (Blood and lymphatic system disorders) | 1
DVT (Blood and lymphatic system disorders) | 1
Neuro decline (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medical Management Plus Apollo MIES (N=50)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Altered mental status (Psychiatric disorders) | 1
Leukocytosis (Blood and lymphatic system disorders) | 2
UTI (Infections and infestations) | 3
Chest pain (General disorders) | 1
Sinus bradycardia (Cardiac disorders) | 2
Hematoma (Blood and lymphatic system disorders) | 1
ICH (Nervous system disorders) | 2
Pneumonia (Infections and infestations) | 3
Atrial fibrillation (Cardiac disorders) | 1
Sepsis (Immune system disorders) | 1
Seizure (Nervous system disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Laryngeal edema (Blood and lymphatic system disorders) | 1
Stroke (Nervous system disorders) | 2
Postoperative hemorrhage (Surgical and medical procedures) | 2
Tremor (Nervous system disorders) | 1
Fever (Infections and infestations) | 2
Desaturation (General disorders) | 1
Pain (General disorders) | 1
Headache (General disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Hiccups (General disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Delusions (Psychiatric disorders) | 1
Hydrocephalus (Nervous system disorders) | 1
Broken Hip (General disorders) | 1
Right shoulder pain (General disorders) | 1
Left hip pain (General disorders) | 1
Amiodarone-induced hypothyroidism (Surgical and medical procedures) | 1
Bowel Perforation (Gastrointestinal disorders) | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1
Tract hemorrhage (Nervous system disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Acute agitation (Psychiatric disorders) | 1
Hypernatremia (Blood and lymphatic system disorders) | 1
Weakness (General disorders) | 1
Syncope (Nervous system disorders) | 1
Dislodged PEG tube (Surgical and medical procedures) | 1
Hypokalemia (Blood and lymphatic system disorders) | 1
Pneumothorax secondary to thoracentisis (Surgical and medical procedures) | 1
Hypertension (Cardiac disorders) | 1
Otomastoiditis (Infections and infestations) | 1
Hyperglycemia (Endocrine disorders) | 1
Thromboembolic event (Blood and lymphatic system disorders) | 1
Wound infection (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-10-24): https://cdn.clinicaltrials.gov/large-docs/15/NCT02654015/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-29): https://cdn.clinicaltrials.gov/large-docs/15/NCT02654015/ICF_001.pdf